## ENHANCING ENGAGEMENT WITH DIGITAL MENTAL HEALTH CARE STUDY00010958

07/03/2024

NCT04507360

Aim 3B Statistical Analysis Plan. For Study 1, all research questions were examined via logistic regressions. We assessed whether participants' first condition (i.e., demographics survey or Next Steps survey) predicted the odds of disengagement. Within participants who completed the demographics survey, we examined whether the odds of disengaging and clicking a featured resource on the screening results page significantly differed for participants in the Tailored Resources to Demographics condition compared to control (i.e., Generic Response + Generic Resources). Within participants from the Next Steps survey condition, we tested whether engagement significantly differed for participants shown Tailored Response + Generic Resources, Generic Response + Tailored Resources to Desired Resources, and Tailored Response + Tailored Resources to Desired Resources compared to control. We aimed to identify the optimal tailoring strategy by comparing engagement across all tailoring conditions, with Tailored Resources to Demographics set as the reference group. For Study 2, research questions were examined via t-tests and Cohen's d effect sizes comparing engagement, short-term restructuring effectiveness, longer-term effectiveness (e.g., skill acquisition, reductions in depression and anxiety), and heterogeneous treatment effects by condition (i.e., control, DIY tool without AI, and DIY tool with AI).